CLINICAL TRIAL: NCT04628845
Title: Evaluation of Endo-perio Lesion's Treatment Using Additional Diode Laser 940nm.
Brief Title: Endo-perio Lesion's Treatment With Using Diode Laser 940nm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Elżbieta Dembowska, Principal Investigator, Pomeranian Medical University Szczecin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Periodontitis; Endodontic Inflammation
Keywords: EPL; periodontitis; laser; CBCT
MeSH Terms: conditions — Periodontitis; Pulpitis | interventions — Lasers

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SRP and endontic treatment without laser 940nm (Placebo Comparator): Periodontal pockets's treatment of scaling, root debridement and endodontic treatment of root canals without using laser 940nm.
  Interventions: Device: Endo-perio therapy without laser 940nm
- SRP and endodontic treatment with laser 940nm (Active Comparator): Periodontal pockets's treatment of scaling, root debridement and endodontic treatment of root canals with using laser 940nm.
  Interventions: Device: Endo-perio therapy with laser 940nm

INTERVENTIONS:
Device: Endo-perio therapy with laser 940nm — Periodontal pockets's treatment of scaling, root debridement and endodontic treatment of root canals with using laser 940nm.
  Arms: SRP and endodontic treatment with laser 940nm
Device: Endo-perio therapy without laser 940nm — Periodontal pockets's treatment of scaling, root debridement and endodontic treatment of root canals
  Arms: SRP and endontic treatment without laser 940nm

SUMMARY:
Periodontal marginal and periapical diseases cause a huge destruction of tissues surrounding the tooth with periodontal patients. Treatment consists on elimination of pathogens, which are presented in periodontal pockets and also in root canals. To increase efficiency of endo-perio treatment there is used diode laser wavelength 940nm. Laser disinfection is done in periodontal pockets and root canals.

The aim of the study is to evaluate the effectiveness of treatment of endo-perio lesions with use of medicaments and diode laser.

The study will present cases of endo-perio lesions around molars in investigated and control group. Teeth were subjected to endodontic and periodontological treatment. The roots and pockets have been disinfected with a diode laser only in investigated group. In the both groups between the visits into root canals there were applied alkaline paste. The treatment was completed after 6 months. Before the beginning and after the end of treatment there were made a two-dimensional image and CBCT. CBCT was subjected to manual segmentation. The resulting streolitographic models were allowed to check the change of bone volume.

DETAILED DESCRIPTION:
This study will presented the cases of two groups of patients, in which the endo-perio lesions were reported. The study protocol was approved by the Institutional Ethics Commission of Pomeranian University (No: KB-0012/29/17). Each subject provided informed consent after explanation of the protocol, risk and benefits of study.The both groups counted the same amount of molar teeth - ten molars in investigated (n=10) and in control group (n=10). In the study there were 9 men and 11 women aged between 35 and 58 years.

The study was performed according to split-teeth design, computerized randomly allocated to the control or the investigated group. At first group (investigated group) there were implemented periodontal and endodontic treatment with additional using diode laser wavelength 940 nm. The same steps were made in control group, however without using diode laser in medical procedures.

The first step was to do the clinical measurements (PD,CAL, tooth mobility, vitality test, occlusal condition) and analysis of pantomographic picture, the patients were diagnosed with third grade periodontitis The depth of periodontal pockets (PD) were checked by using manual periodontal probe (UNC 15, Hu-Friedy) on six sites. The classified teeth, which were diagnosed perio-endo lesions, were showed any vitality during testing faradic and ethyl chloride. The teeth did not respond properly. Also the tested teeth were checked with using Periotest M (Medizintechnik Gulden) in both groups before and after the treatment.

Every enrolled patients were checked by using the T-scan Novus (Tekscan). T-scan system records patients bite force, dynamics, including occlusal force, location and timing.

The treatment in EPL should be carried out in two ways- periodontal and endodontic. One of these ways there is mechanical non-surgical treatment of periodontium and endodontic way is eliminated the bacteria, which inside in root canals.

ELIGIBILITY:
Inclusion Criteria:

* advanced periodontitis stage III, with endo-periodontal lesion without root damage,
* presence of at least 20 teeth,
* at least one molar tooth in each quadrant with a minimum of four teeth.

Exclusion Criteria:

-systemic illnesses (unbalanced diabetes mellitus, immunosuppressive drug or HIV), -

* pregnancy or lactation,
* smoking or alcoholism.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-08-31 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
PD | up to 3 months
  periodontal pocket depht
Mobility Tooth | up to 6 months
  checking mobility with using Periotest
CBCT and STL | up to 6 months
  Cone Bean Computed Tomography, stereolithographic models

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Homik-Rodzińska, Msc, Study Director — lek.dent. Aleksandra Homik-Rodzińska
Locations (1):
- Pomeranian Medical University, Szczecin, West Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Documentation of study participants in paper form will be kept at the Department of Periodontology. We provide information on aggregate results in tables and statistical analysis after contact by email.